CLINICAL TRIAL: NCT02368821
Title: From Cytotrophoblast to Syncytiotrophoblast - Telomere Length, Aggregate Formation and Senescence in Placenta From Complicated Pregnancies Compare to Placenta From Normal Pregnancies.
Brief Title: From Cytotrophoblast to Syncytiotrophoblast
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0202-14-MMC
Record Dates: First submitted 2015-01-15; First posted 2015-02-23 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-01

CONDITIONS: Syncytiotrophoblast
Keywords: cytotrophoblast; syncytiotrophoblast; placentas; intrauterine growth restriction; preeclampsia; placenta accrete
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — paraffin blocks placenta cell cultures
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal pregnancy: placental from normal pregnancy
- complacted pregnancy: placental from complicated pregnancy ( intrauterine growth restriction, preeclampsia , placenta accrete

SUMMARY:
A deeper understanding of the syncytiotrophoblast development processes and its properties may allow a better understanding of the placenta pathological process for the development of treatment models for the relevant pregnancy complications.The aim of this study is to compare telomere length, aggregate formation, and senescence markers in placentas from complicated pregnancy with placentas from normal pregnancy.

DETAILED DESCRIPTION:
Protocol summary No. 2 for research 0202-14 of date: 22/11/2014. Rationale for the research A deeper understanding of the syncytiotrophoblast development processes and its properties may allow a better understanding of the placenta pathological process for the development of treatment models for the relevant pregnancy complications.

The aim of this study is to compare telomere length, aggregate formation, and senescence markers in the syncytiotrophoblast of placentas from complicated pregnancy with placentas from normal pregnancy.

Telomere lenght and aggregate formation will be assessed by the fluorescent intensity of telomere FISH.

Senescence will be assessed by immunohistochemistry for the markers - SAHF, cyclin dependent kinase inhibitors p16/p21, HLAX, ERVWE1, SA-B-gal.

The study groups

1. A retrospective arm - paraffin blocks which were collected over the years from placentas from complicated pregnancy ( intrauterine growth restriction, preeclampsia , placenta accrete) will be compared to blocks of placentas from normal pregnancies.
2. The prospective arm - placental from complicated pregnancy ( intrauterine growth restriction, preeclampsia , placenta accrete) . Will be compared to placentas of normal pregnancies.
3. A laboratory model based on human placenta cell cultures

ELIGIBILITY:
Inclusion Criteria:

* placentas from normal and complicated pregnancy

Exclusion Criteria:

* women consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: placentas from normal and complicated pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Length of telomere and senescence markers amount in the placentas. | 2 years